CLINICAL TRIAL: NCT01663935
Title: Interventional Study of Levodopa Replacement on Retinal Function in Oculocutaneous Albinism
Brief Title: Vision Response to Dopamine Replacement
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-1576; 2012-0023 (Other: Study team)
Record Dates: First submitted 2012-08-09; First posted 2012-08-14 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Albinism; Oculocutaneous Albinism
Keywords: levodopa; Albinism; dopamine; oculocutaneous albinism; vision; retina function
MeSH Terms: conditions — Albinism; Albinism, Oculocutaneous | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levodopa/carbidopa 4mg/kg/day (Other): Treatment drug taken orally three times daily
  Interventions: Drug: Levodopa/carbidopa

INTERVENTIONS:
Drug: Levodopa/carbidopa — This study will have an intent to treat goal. Anyone that fits the inclusion criteria for the study will be entered and receive study drug.
  Other Names: Sinemet; Atamet; Parcopa

SUMMARY:
The purpose of the study is to evaluate and document physiologic and functional changes in visual performance and retinal function of patients diagnosed with albinism (a dopamine deficiency state) following a trial of oral Levodopa/carbidopa treatment.

DETAILED DESCRIPTION:
In this study the investigators propose that the retina itself in albinism is deficient in dopamine, and vision improvement will occur as a result of improved retinal function in response to the deficient neurotransmitter dopamine. This study has a pretest-posttest design in order to determine if improvement in vision is in response to replacement of deficiency (dopamine). The electroretinography (ERG) testing and optical coherence tomography (OCT) will be critical determinants to confirm vision improvement as a result of improved retinal function, but are not primary outcome data. Main outcome measures will be collected at pre-treatment, 1 month, 3 months, and 4 months. Change in visual acuity as measured in logMAR by Snellen or sweep visual evoked potential (SVEP) after 3 months of treatment is the primary outcome. Patients include OCA1a patients, OCA1b, OCA2, and unclassified Oculocutaneous albinism (OCA). OCA1a patients clinically are known to have the worst vision, and physiologically have the lowest (or absent) levels of tyrosinase function (Dopamine Production). All patients will be treated with Levodopa/carbidopa 4mg/kg/day in three divided doses.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of oculocutaneous albinism
* age over 3 and weight over 25 lbs.

Exclusion Criteria:

* ocular only albinism
* ocular pathology other than albinism
* neurologic disease, history of myocardial infarction, history of clinical depression, pregnancy

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10-17 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Struck, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Levodopa/Carbidopa 4mg/kg/Day
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Levodopa/Carbidopa 4mg/kg/Day
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Non hispanic or latino/ white | 16
  Race/Ethnicity: non hispanic or latino/ asian | 3
  Race/Ethnicity: hispanic or latino | 1
Region of Enrollment [Number; unit: participants]
  United States | 19
  Canada | 1

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity Change
Description: Change in visual acuity from baseline to 3 months as measured in logMAR by Snellen or Sweep visual evoked potential (SVEP). logMar lower values equals better visual outcome.
Time Frame: 3 months
Population: participants pre and post treatment per protocol
Measure: Mean (Standard Deviation); unit: logMar
Arm/Group | Levodopa/Carbidopa 4mg/kg/Day
Number analyzed (Participants) | 19
logMar | .774 (.207)

2. Other Pre Specified Outcome: Contrast Sensitivity
Description: Ancillary testing of visual/retinal function with contrast sensitivity testing. Contrast sensitivity testing measures how well the eyes can distinguish between finer and finer light increments compared to dark. This test is a chart with different capital letters organized in horizontal lines. The contrast decreases with each line. The person will move down the chart to determine the least level of contrast they can see.
Time Frame: 3 months
Population: participants pre and post medication per protocol for contrast sensitivity. Range could be anywhere from a score of 0 to 75 for each eye. The higher the score the more letters they could see in low contrast.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Levodopa/Carbidopa 4mg/kg/Day
Number analyzed (Participants) | 19
Number analyzed (eyes) | 38
score on a scale | 23.7 (21.6)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each patient starting at baseline through the month 4 study follow up visit.
Arm/Group | Levodopa/Carbidopa 4mg/kg/Day
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/35/NCT01663935/Prot_SAP_000.pdf